CLINICAL TRIAL: NCT02247934
Title: Development of a Patient-Reported Outcome Measure to Assess Symptoms in Patients With Primary Sclerosing Cholangitis (PSC)
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: A-13601-000
Record Dates: First submitted 2014-09-05; First posted 2014-09-25 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary sclerosing cholangitis; PSC
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concept elicitation interviews (Step I): Approximately 20 participants will be included.
- Cognitive interviews (Step II): Approximately 30 participants will be included.

SUMMARY:
The objectives of this qualitative study are to elicit concepts about symptoms that are important to patients with primary sclerosing cholangitis (PSC), as well as the key impacts of symptoms on patients' day-to-day functioning.

DETAILED DESCRIPTION:
In Step I, concept elicitation one-on-one interviews (via telephone or in person) will be conducted. The aims of the concept elicitation interviews are to:

1. Identify the most common symptoms, as well as the most important symptoms, for patients with PSC, and
2. Assess whether these symptoms impact day-to-day functioning

An instrument will be developed based on the symptoms reported and in Step II of the study, the performance of the instrument will be assessed with further interviews.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PSC based on liver biopsy or diagnostic imaging, with diagnosis made at least three months prior to screening
* Patient report of PSC symptoms associated with PSC diagnosis
* Able to speak, read, and understand English
* Willing and able to provide written informed consent to participate in the research study

Exclusion Criteria:

* Patients with other causes of liver or biliary disease, including viral hepatitis, alcoholic liver disease, primary biliary cirrhosis, and secondary sclerosing cholangitis
* Patient with history of liver cirrhosis
* Patients with history of cholangiocarcinoma
* Patients who have received a liver transplant
* Patients currently enrolled in PSC clinical trials; and
* STEP II ONLY: Enrolled in or participated in Step I of this study (concept elicitation)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from approximately 5 clinical sites based in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
List Primary Sclerosing Cholangitis (PSC) Symptoms for inclusion in patient questionnaire | Up to 12 months
  Interview participants to generate a list of the most common symptoms, as well as the most important symptoms, experienced by patients with PSC, and whether each symptom impacts day-to-day functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Myers, MD, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - University of Colorado Hospital, Denver Health Medical Center, Aurora, Colorado
  - University of Miami Miller School of Medicine - Schiff Center for Liver Diseases, Miami, Florida
  - Evidera, Bethesda, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Organ Care Research Swedish Medical Center, Seattle, Washington